CLINICAL TRIAL: NCT04118205
Title: REtinaL Imaging & Ambulatory BLood PrEssure: Validating Ultra-widefield Retinal Imaging Derived Biomarkers Against Ambulatory Blood Pressure
Brief Title: REtinaL Imaging & Ambulatory BLood PrEssure
Acronym: RELIABLE
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Optos, PLC (Industry); NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC18080
Record Dates: First submitted 2019-10-01; First posted 2019-10-08 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High blood pressure is a common condition which generally does not have any symptoms. Its estimated that around one third of people with high blood pressure do not know they have it. The back of the eye called the retina is one of the few places in the human body allowing easy observation of blood vessels. This study aims to see if simple non-invasive imaging of the blood vessels of the retina will highlight people with high blood pressure.

DETAILED DESCRIPTION:
This will be a prospective, single centre study recruiting patients who are attending the ambulatory blood pressure clinic at the Western General Hospital. Suitable patients will be approached, and if they consent will have pictures of the back of each of their eyes taken. These pictures will then be reviewed, with certain measurements taken of the small blood vessels which can been seen at the back of the eye. These measurements will then be compared to the participants blood pressure readings to see if they might accurately correlate to blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Attending ambulatory blood pressure clinic
* Able to undertake ambulatory BP measurement
* Able to undertake single clinic-based BP measurement
* Able to undergo UWF retinal imaging with a SLO
* Aged 18 to 90
* Able to give informed consent

Exclusion Criteria:

* People with known history of retinal surgery
* People under the age of 18 years.
* People that cannot: manoeuvre themselves to the SLO unaided, sit upright in a chair or wheelchair or position themselves comfortably for imaging.
* People with epilepsy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants attending a hypertensive clinic at the Western General Hospital in Edinburgh will be asked to consent to ultra-wide field retinal imaging, subject to the inclusion and exclusion criteria below. It is expected that between 25 and 50 participants per week attend the clinic, of which approximately 50% are attending without a known diagnosis of hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Does retinal arteriovenous ratio correlate to systolic blood pressure | 1 day
  Retinal arteriovenous ratio (as measured by ultra-wide field imaging) will be correlated to mean daytime systolic blood pressure (as measured by 24-hour ambulatory blood pressure monitoring)

SECONDARY OUTCOMES:
Does retinal arteriovenous ratio correlate to clinic systolic blood pressure | 1 day
  Retinal arteriovenous ratio (as measured by ultra-wide field imaging) will be correlated to clinic systolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, City Of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT04118205/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04118205/SAP_001.pdf